CLINICAL TRIAL: NCT03043560
Title: Developing Neuronal KCNQ Channel Modulators for Mood Disorders
Brief Title: Study to Treat Major Depressive Disorder With a New Medication
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: James Murrough (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, James Murrough, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: GCO 16-0374; 1R61MH111932-01 (NIH)
Record Dates: First submitted 2017-02-02; First posted 2017-02-06 (Estimated); Results first posted 2020-10-23 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-09

CONDITIONS: Depressive Disorder; Anhedonia
Keywords: depression; anhedonia; reward
MeSH Terms: conditions — Depressive Disorder; Anhedonia; Depression | interventions — ezogabine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ezogabine (Experimental): Participants will receive treatment with ezogabine up to 900mg/day.
  Interventions: Drug: Ezogabine
- Placebo (Placebo Comparator): Participants will receive treatment with a matching placebo pill.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Ezogabine — daily for 5 weeks
  Other Names: Potiga
  Arms: Ezogabine
Drug: Placebos — placebo pill daily for 5 weeks
  Arms: Placebo

SUMMARY:
This project is designed to examine the neuronal KCNQ2/3 potassium (K+) channel subtype as a novel treatment target for mood disorders through the administration of the KCNQ-selective channel opener ezogabine (Potiga, GlaxoSmithKline; FDA-approved for the treatment of seizure disorders).

DETAILED DESCRIPTION:
Depressive disorders are among the most disabling medical conditions worldwide and currently available treatments fall short of addressing this large public health burden. Dysfunction within the brain reward system is emerging as a core feature of depressive disorders, in particular related to deficits in motivation, interest, and response to pleasure (e.g., anhedonia: markedly diminished response to pleasure). Evidences from a series of preclinical studies from our group highlighted the KCNQ subtype of neuronal potassium (K+) channel as a novel target for the treatment of depressive disorders and our human pilot study showed a reduction in anhedonia and related symptoms, and an increased brain response to reward (as measured by functional magnetic resonance imaging [fMRI]) following treatment with ezogabine. Building on this data, the current project will assess reward circuit activity following treatment with ezogabine in depressed patients with a current depressive disorder (Major depressive disorder [MDD], persistent depressive disorder, other specified depressive disorder) and anhedonia (defined by a score ≥ 20 on the Snaith-Hamilton Pleasure Scale [SHAPS]), using fMRI to investigate the cortico-striatal circuit to reward.

This study represents the first part of the R61/R33 National Institutes of Health (NIH) founded project. A clear increase in reward circuit activation in at least one ezogabine treatment group compared to placebo, given acceptable tolerability, will constitute a "go" and the project will move to the next phase (R33), where we aim to examine the relationship between treatment, reward circuit activity, and behavioral and clinical outcomes in a larger, confirmatory efficacy trial of ezogabine for depression with anhedonia.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained from subject and ability for subject to comply with the requirements of the study;
* Men and women, age 18-65;
* Participants must meet DSM-V criteria for current depressive disorder (major depressive disorder [MDD], persistent depressive disorder, other specified depressive disorder) as determined by a study psychiatrist and confirmed using the Structured Clinical Interview for DSM-V (SCID);
* Clinically significant anhedonia as determined by a SHAPS score ≥ 20 at screening;
* Current illness severity is at least moderate, defined as a score of ≥4 on the Clinical Global Impression-Severity (CGI-S) Scale;
* If female of childbearing potential, must agree to use of a medically accepted form of contraception, or else agree to abstinence.

Exclusion Criteria:

* A primary psychiatric diagnosis other than a depressive disorder as defined by DSM-V [co-morbid anxiety disorders (including agoraphobia, generalized anxiety disorder, social anxiety disorder and panic disorder) and Posttraumatic Stress Disorder (PTSD) are allowed] or major cognitive disorder;
* Meets criteria for a substance or alcohol use disorder in the past 6 months;
* Female participants who are pregnant, breastfeeding, or may become pregnant, or unwilling to practice birth control during participation in the study;
* Positive urine toxicology screen for drugs of abuse at the time of screening;
* Any unstable medical illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including ischemic heart disease), endocrinologic, neurologic, immunologic, or hematologic disease;
* Clinically significant abnormalities of laboratory tests, physical examination, or ECG;
* Prolonged QT Interval at screening, operationalized as a QTc of > 480 ms;
* A history of retinal abnormalities (i.e., pigment changes, retinal dystrophy) or findings of retinal pathology on ophthalmological exam at baseline;
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data;
* Use of any dis-allowed medication according to the study protocol;
* Serious and imminent risk of self harm or violence as determined by the PI;
* Extreme illness severity as defined by a GCI-S score >6;
* Any contraindication to MRI including claustrophobia, any trauma or surgery which may have left magnetic material in the body, magnetic implants or pacemakers, and inability to lie still for 1 hour or more;
* History of non-response to electroconvulsive therapy in the current depressive episode

  * Exceptions:

    1. Subjects with a positive urine drug screen for cannabinoids, barbiturates, opiates, amphetamines, or benzodiazepines may be allowed in the study provided that the drug was used for a documented, legitimate medical purpose and/or the use of such products may be discontinued (documented by a negative repeat test) prior to randomization;
    2. Medically appropriate episodic use (up to 3 days) of narcotic analgesics for acute medical indications is allowed (Discussion with PI required)

       * Potential participants will not be discontinued from medication for the purposes of this study. If a patient is taking a protocol dis-allowed medication at the time of screening, the patient may discontinue the medication under the supervision of the treating physician in the case that the patient is not benefiting from the medication or otherwise wishes to discontinue the medication. In no case will a dis-allowed medication be discontinued for the purpose of study participation if the patient is receiving clinical benefit from the medication.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data from this study may be submitted to the National Database for Clinical Research Related to Mental Illness (NDCT). NDCT isa data repository run by the National Institute of Mental Health (NIMH) that allows researchers studying mental illness to collect and share deidentified information with each other. During and after the study, the researchers will send deidentified information about health and behavior and in some cases, genetic information, to NDCT. Other researchers nationwide can then file an application with the NIMH to obtain access to deidentified study data for research purposes.

REFERENCES:
- [Derived] Costi S, Morris LS, Kirkwood KA, Hoch M, Corniquel M, Vo-Le B, Iqbal T, Chadha N, Pizzagalli DA, Whitton A, Bevilacqua L, Jha MK, Ursu S, Swann AC, Collins KA, Salas R, Bagiella E, Parides MK, Stern ER, Iosifescu DV, Han MH, Mathew SJ, Murrough JW. Impact of the KCNQ2/3 Channel Opener Ezogabine on Reward Circuit Activity and Clinical Symptoms in Depression: Results From a Randomized Controlled Trial. Am J Psychiatry. 2021 May 1;178(5):437-446. doi: 10.1176/appi.ajp.2020.20050653. Epub 2021 Mar 3. PMID 33653118

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from Sept 2017 through August 2019
Groups:
- Ezogabine: Ezogabine up to 900mg/day daily for 5 weeks
- Placebo: Matching placebo pill daily for 5 weeks
Period: Overall Study
Arm/Group | Ezogabine | Placebo
Started | 21 | 24
Completed | 20 | 21
Not Completed | 1 | 3
Not completed — Discontinued Intervention | 1 | 2
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ezogabine | Placebo | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (13.6) | 38.9 (14.3) | 41.5 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 11 | 12 | 23
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — as reported by the study participant
  Participants
    White/Caucasian | 12 | 12 | 24
    Black/African American | 5 | 7 | 12
    Hispanic/Latino | 6 | 9 | 15
Employment at least Part-Time [Count of Participants; unit: Participants] | 9 | 14 | 23
Educational Attainment - ast least some college [Count of Participants; unit: Participants] | 15 | 21 | 36
Relationship Status - Single, Never Married [Count of Participants; unit: Participants] | 8 | 13 | 21
Primary Diagnosis [Count of Participants; unit: Participants]
  Major Depressive Disorder | 21 | 23 | 44
  Persistent Depressive Disorder | 0 | 1 | 1
Current Major Depressive Episode [Count of Participants; unit: Participants] | 21 | 22 | 43
Age at Onset of Depression [Mean (Standard Deviation); unit: years] | 28.3 (15.6) | 21.7 (11.5) | 24.3 (14.0)
Current Depressive Episode Duration [Median (Inter-Quartile Range); unit: months] | 72 [6 to 180] | 24 [9.5 to 54] | 30 [10 to 120]
Generalized Anxiety Disorder [Count of Participants; unit: Participants] | 11 | 10 | 21
Posttraumatic Stress Disorder (PTSD) [Count of Participants; unit: Participants] | 4 | 8 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in Ventral Striatum (VS) Activation
Description: change in activation during reward anticipation within the bilateral VS from baseline (Study Visit 0) to the primary outcome visit (Study Visit 5) as measured by functional MRI during the incentive flanker task (IFT). The IFT, like the Monetary Incentive Delay task, permits discrete modeling of brain activity during anticipation of an incentive.
  Functional scans were preprocessed and denoised for motion and physiological noise using multi-echo independent component analysis (ME-ICA). Task-based modeling was conducted using AFNI and FSL software. The primary outcome for reward anticipation was the contrast of reward cue compared to neutral cue (reward>neutral cue). The primary imaging outcome was analyzed using a linear mixed model with a single random intercept term treating time as discrete or continuous as appropriate.
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: Bold Oxygen-level Dependent (BOLD) Signa
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
Bold Oxygen-level Dependent (BOLD) Signa
  baseline | -0.26 (0.69) | 0.95 (0.79)
  5 weeks | 0.176 (0.81) | 0.015 (0.68)

2. Secondary Outcome: Change in Snaith-Hamilton Pleasure Scale (SHAPS)
Description: The SHAPS is a well-validated 14-item self-report questionnaire commonly used to assess anhedonia. Each item on the SHAPS is worded so that higher scores indicate greater pleasure capacity. A total score can be derived by summing the responses to each item. Items answered with "strongly agree" are coded as "1", while a "strongly disagree" response was assigned a score of "4." Total scores on the SHAPS can range from 14 to 56, with higher scores corresponding to higher levels of anhedonia.
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  Baseline | 38.7 (8.1) | 33.7 (6)
  5 weeks | 27.5 (8.5) | 30 (10.9)

3. Secondary Outcome: Clinical Global Impression - Improvement (CGI-I)
Description: A widely administered clinician rated global measure of the degree of improvement from the initial assessment in subject overall illness severity. 7 point scale rated as: 1, very much improved; 2, much improved; 3, minimally improved; 4, no change; 5, minimally worse; 6, much worse; or 7, very much worse.
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  baseline | 4 (0.2) | 4 (0.4)
  5 weeks | 2.1 (1) | 2.8 (1.3)

4. Secondary Outcome: Clinical Global Impression - Severity (CGI-S)
Description: Clinician rated global measure of subject overall illness severity. a 7-point scale rated as 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  baseline | 4.4 (0.5) | 4.6 (0.6)
  5 weeks | 2.6 (1.2) | 3.3 (1.2)

5. Secondary Outcome: Anticipatory and Consummatory Interpersonal Pleasure Scale (ACIPS)
Description: A measure specifically designed to assess hedonic capacity for social and interpersonal pleasure.The ACIPS is a 17-item self-report measure scored on a likert scale, ranging from 1 (very false for me) to 6 (very true for me). Full scale from 17-102, higher score indicates higher hedonic capacity
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  baseline | 46.1 (15.1) | 53.7 (15)
  5 weeks | 65.1 (22.8) | 59 (23.5)

6. Secondary Outcome: Montgomery-Asberg Depression Rating Scale (MADRS)
Description: A 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each items is scored 0 (normal) to 6 (severe depression) with overall score ranges from 0 (normal) to 60 (severe depression).
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  baseline | 28.3 (6.1) | 26.8 (5.1)
  5 weeks | 12.7 (8.7) | 18.5 (10.1)

7. Secondary Outcome: World Health Organization Disability Assessment Schedule 2.0 (WHODAS 2.0)
Description: A 12-item generic assessment instrument that measures the level of functioning. Each item is scored from 0 to 4 and the items are summed to provide a total score. The score therefore ranges from 0 to 48, with higher scores indicating greater disability.
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  baseline | 15.5 (7.5) | 16.5 (9.4)
  5 weeks | 10.2 (9.5) | 11.6 (9.8)

8. Secondary Outcome: Temporal Experience of Pleasure Scale (TEPS)
Description: The TEPS is composed of 18-items rated on a likert-type scale ranging from 1 (Very True for me) to 6 (Very False for me), and yields two subscales. Ten items make up the TEPS-Anticipatory Pleasure (TEPS-ANT) scale with a range from 10 (not motivated) to 60 (highly motivated). The other eight TEPS items make up the TEPS-Consummatory Pleasure (TEPS-CON) scale; range from 8 (not responsive) to 48 (highly responsive). Total scores range is 18-108. Lower scores indicate greater levels of anhedonia.
Time Frame: baseline and 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  TEPS-ANT baseline | 26.3 (8.3) | 28.6 (8.7)
  TEPS-ANT 5 weeks | 37.3 (10.5) | 32.4 (11.5)
  TEPS-CON baseline | 24.8 (8.1) | 25.6 (7.6)
  TEPS-CON 5 weeks | 32.2 (6) | 29.9 (10.5)

9. Secondary Outcome: Specific Loss of Interest and Pleasure Scale (SLIPS)
Description: The SLIPS is a recently developed and validated measure of anhedonia that is tailored to detect recent changes in anhedonia. A 23-item measure, each item range from 0-3. Full scale from 0 to 69, higher score indicates more recent changes.
Time Frame: baseline 5 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Ezogabine | Placebo
Number analyzed (Participants) | 21 | 24
score on a scale
  baseline | 32.3 (9.8) | 28.8 (10.4)
  5 weeks | 16.3 (16.7) | 21.5 (16.8)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Ezogabine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 21/21 | 19/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ezogabine (N=21) | Placebo (N=24)
Abdominal Pain (Gastrointestinal disorders) | 2 | 3
Anxiety (Psychiatric disorders) | 1 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 1
Disturbance in attention (Nervous system disorders) | 3 | 0
Dizziness (Nervous system disorders) | 21 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 7
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Memory impairment (Nervous system disorders) | 1 | 2
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 3 | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Panic attack (Psychiatric disorders) | 2 | 0
Polyuria (Renal and urinary disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Restlessness (Psychiatric disorders) | 0 | 1
Sedation (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 2 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Vision blurred (Eye disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 2 | 1
Other (General disorders) | 9 | 8

LIMITATIONS AND CAVEATS:
The relatively small sample size and termination of enrollment prior to the planned target limit conclusions regarding efficacy and generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-06-01): https://cdn.clinicaltrials.gov/large-docs/60/NCT03043560/SAP_000.pdf
  • Study Protocol (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/60/NCT03043560/Prot_001.pdf